CLINICAL TRIAL: NCT00260026
Title: Safety and Pharmacokinetic Study of Jin Fu Kang In Combination With Docetaxel for Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: Safety and Pharmacokinetics of Jin Fu Kang in Comb w/Docetaxel for Patients w/Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-010
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel
Drug: Jin Fu Kang

SUMMARY:
Researchers from Memorial Sloan-Kettering Cancer Center are conducting a research study on a Chinese herbal medicine known as "Jin Fu Kang". We want to see if this can help patients with advanced lung cancer. Jin Fu Kang might reduce the growth of cancer or improve quality of life. You are eligible for this trial because your cancer has progressed after prior chemotherapy and your doctor has recommended further chemotherapy treatment.

Lung cancer that has been confirmed and that has spread is called advanced cancer. There is no known permanent cure for advanced lung cancer, but chemotherapy may temporarily shrink the cancer and improve the quality of patients' lives.

DETAILED DESCRIPTION:
Jin Fu Kang is a herbal medicine specially developed in China for the treatment of lung cancer. It is based on a traditional medicine that is widely used and appears to be safe. Although clinical trials in China suggest that Jin Fu Kang may be of benefit, it has never been researched in patients with lung cancer in the United States. As such, its risks and benefits are not fully understood.

The scientific aims are to determine the toxicity of Jin Fu Kang/docetaxel combination treatment in patients with non-small cell lung cancer, to determine whether Jin Fu Kang alters the pharmacokinetics of docetaxel and to provide preliminary efficacy and survival data for Jin Fu Kang/docetaxel combination treatment in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

-Patients must meet all of the following inclusion criteria:

* Pathologic confirmation of stage III or IV NSCLC.
* Docetaxel therapy for cancer is clinically indicated.
* KPS>=60% *ANC<1,000/mcl and Platelets<100/mcl

Exclusion Criteria:

-Patients must meet none of the following exclusion criteria:

* WBC< 4,000/µl, hemoglobin < 10 g/dl, platelet count < 100,000/µl, total bilirubin > ULN, AST >1.5 x ULN, alkaline phosphatase > 2.5 x ULN, creatinine > 1.5 mg/dl or creatinine clearance < 50 ml/min/1.7 m2), (ANC > 10,000/µl)
* Prior docetaxel
* Patient must have recovered from all previous treatment-related toxicity
* Concurrent use of any botanicals for anticancer intent
* Use of Jin Fu Kang or any of its constituent botanicals in the previous three weeks.
* History of allergy to any of the constituent botanicals in Jin Fu Kang.
* Pregnant or lactating women or women of childbearing potential not using effective contraception. A negative pregnancy test must be documented during the screening period for women of childbearing potential.
* Concurrent active cancer.
* Concurrent use of immunosuppressives: as an immunostimulant, astragalus-containing products are contraindicated for patients on immunosuppressive therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-11; Study Completion 2007-01

PRIMARY OUTCOMES:
To determine the toxicity of Jin Fu Kang / docetaxel combination treatment in patients with previously treated non-small cell lung cancer.

SECONDARY OUTCOMES:
To determine whether Jin Fu Kang alters the pharmacokinetics of docetaxel.
To provide preliminary efficacy and survival data for Jin Fu Kang / docetaxel combination treatment in patients with previously treated non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer A Rizvi, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org